CLINICAL TRIAL: NCT03315104
Title: A Randomized, Double-Blind, Placebo-Controlled Dose Ranging Study Evaluating Safety, Pharmacokinetics and Clinical Benefit of FLU-IGIV in Hospitalized Patients With Serious Influenza A Infection
Brief Title: Exploring Safety & Clinical Benefit of Anti-Influenza Immunoglobulin Intravenous in Hospitalized Adults With Influenza A
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emergent BioSolutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IA-001
Record Dates: First submitted 2017-10-06; First posted 2017-10-19 (Actual); Results first posted 2020-10-05 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Influenza A H3N2; Influenza A H1N1
Keywords: influenza A; hospitalized; H1N1; H3N2; human flu; respiratory tract infection; serious illness; flu
MeSH Terms: conditions — Orthomyxoviridae Infections; Influenza, Human; Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: Staggered enrollment for the first 9 subjects, then parallel low and high dose treatment with a placebo group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- FLU-IGIV High Dose (Experimental): Participants will receive a single infusion of high dose of FLU-IGIV, administered over approximately 3 hours on Day 1. Participants will also receive standard of care (SOC) antiviral treatment for flu. Administered intravenously at a dose of 450 mL of 65 g/mL FLU-IGIV diluted to 500 mL with normal saline. Participants also received standard of care (SOC) antiviral treatment for flu.
  FLU-IGIV: Single dose, sterile liquid formulation for IV administration.
  Interventions: Biological: FLU-IGIV
- FLU-IGIV Low Dose (Experimental): Participants will receive a single infusion of low dose of FLU-IGIV, administered over approximately 3 hours on Day 1. Participants will also receive SOC antiviral treatment for flu. Administered intravenously at a dose of 225 mL of 65 g/mL FLU-IGIV diluted to 500 mL with normal saline. Participants also received standard of care (SOC) antiviral treatment for flu.
  FLU-IGIV: Single dose, sterile liquid formulation for IV administration.
  Interventions: Biological: FLU-IGIV
- FLU-IGIV Placebo (Placebo Comparator): Participants will receive a single infusion of placebo for FLU-IGIV, administered over approximately 3 hours on Day 1. Participants will also receive SOC antiviral treatment for flu. Administered IV as 500 mL of normal saline. Participants also received standard of care (SOC) antiviral treatment for flu.
  Placebo for FLU-IGIV: Single dose, normal saline solution for IV administration.
  Interventions: Other: Placebo for FLU-IGIV

INTERVENTIONS:
Biological: FLU-IGIV — Single dose, sterile liquid formulation for IV administration.
  Other Names: Anti-influenza immunoglobulin intravenous (Human); NP-025
  Arms: FLU-IGIV High Dose; FLU-IGIV Low Dose
Other: Placebo for FLU-IGIV — Single dose, normal saline solution for IV administration.
  Arms: FLU-IGIV Placebo

SUMMARY:
Influenza, or the flu, is an infectious respiratory disease that can range in severity from mild to severe to even death. This study aims to evaluate a treatment for people who are hospitalized with the flu. The study is looking to see if antibodies collected from people who have recovered from the seasonal flu or who have had the seasonal flu shot can be used safely as a study drug to treat hospitalized patients with severe flu infections. Also, this study will help to find the right dose for this study drug for treatment of severe flu in hospitalized patients. Overall, this study will evaluate if the hospitalized patients receiving standard of care along with the study drug get better more quickly than those treated with standard of care and placebo. The study drug that contains antibodies against the flu is called anti-influenza immunoglobulin intravenous (FLU-IGIV).

ELIGIBILITY:
Inclusion Criteria:

* Provision of voluntary informed consent in writing by patient, or legally authorized representative.
* Age ≥ 18 years of age.
* Locally determined positive influenza A infection (Rapid Antigen (Ag) Test or PCR) from a specimen obtained within 2 days prior to randomization.
* Onset of symptoms ≤ 6 days before randomization, defined as when the patient first experienced at least one respiratory symptom or fever.
* Hospitalized (or in observation unit) with influenza, with anticipated hospitalization for more than 24 hours and will be/already are receiving antiviral SOC.
* Experiencing ≥ 1 respiratory symptom (ex. cough, sore throat, nasal congestion) and ≥ 1 constitutional symptom (ex. headache, myalgia, feverishness or fatigue).
* For women of child-bearing potential: willingness to abstain from sexual intercourse or use at least 1 form of hormonal or barrier contraception through Day 60 of the study.
* Willingness to have blood and respiratory samples obtained and stored.
* National Early Warning Score (NEW score) ≥ 3 at screening.

Exclusion Criteria:

* Use of any investigational product within the past 30 days prior to screening.
* History of hypersensitivity to blood or plasma products (as judged by the site investigator).
* History of allergy to latex or rubber.
* Known medical history of IgA deficiency.
* Pregnancy or lactation.
* Medical conditions for which receipt of a 500 mL volume of intravenous fluid may be dangerous to the patient (e.g. decompensated congestive heart failure), based on investigator's medical opinion with careful consideration of lab results.
* Liver function: liver function test (LFT) > 2.5 times upper limit of normal (ULN).
* Renal Function: glomerular filtration rate (GFR) < 60 mL/min/1.73 m2 (age and sex adjusted).
* A pre-existing condition or use of a medication that, in the opinion of the site investigator, may place the individual at a substantially increased risk of thrombosis (e.g. cryoglobulinemia, severe refractory hypertriglyceridemia, or clinically significant monoclonal gammopathy).
* An opinion of the investigator that it would be unwise to allow participation of the patient in the study (the reason for exclusion of the patient must be documented).
* Receiving extracorporeal membrane oxygenation (ECMO).
* Anticipated life expectancy of < 90 days.
* Confirmed bacterial pneumonia or any concurrent respiratory viral infection that is not influenza A (ex. respiratory syncytial virus (RSV) infection).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2019-06-17 (Actual); Study Completion 2019-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Hall, Study Director — Emergent BioSolutions Inc
Locations (55):
- United States (42):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - HonorHealth, Scottsdale, Arizona
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - University of California, Irvine Emergency Medicine, Orange, California
  - Denver public Health, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Christiana Care Health Systems, Newark, Delaware
  - Northside Hospital, Atlanta, Georgia
  - Atlanta Institute for Medical Research Inc., Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Kansas medical Center, Kansas City, Kansas
  - John Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Wayne State University/Detroit Receiving Hospital, Detroit, Michigan
  - Wayne State University/Sinai Grace Hospital, Detroit, Michigan
  - Providence-Providence Park Hospital, Southfield, Southfield, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Pulmonlx LLC Pulmonary & Critical Care Medicine, Greensboro, North Carolina
  - Premier Health Miami Valley Hospital, Dayton, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - St Luke's University Health Network, Bethlehem, Pennsylvania
  - Einstein Medical Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Regional Health, Rapid City, South Dakota
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Michael E. DeBakey VA Medical Center, Houston, Texas
  - UT Health San Antonio, San Antonio, Texas
  - University of Utah HealthCare, Salt Lake City, Utah
  - Carilion Medical Center, Roanoke, Virginia
  - MultiCare Institute for Research & Innovation, Tacoma, Washington
- Canada (6):
  - Foothills Medical Centre, Calgary, Alberta
  - Health Sciences Center, Winnipeg, Manitoba
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Grace Hospital, Winnipeg, Manitoba
  - CISSS BSL/Hopital Regional de Rimouski, Rimouski, Quebec
  - Ciusss McQ, Trois-Rivières, Quebec
- Puerto Rico (2):
  - Mayaguez Medical Center, Mayagüez
  - San Cristobal Hospital, Ponce
- Spain (5):
  - Hospital Clinic of Barcelona, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitari Mutua Terrassa, Barcelona
  - Reina Sofia University Hospital, Córdoba
  - Hospital Universitari de Tarragona Joan XXIII, Tarragona

IPD SHARING:
Plan to Share IPD: Yes
Post results and upload the supporting information.
Supporting Information: Study Protocol, SAP
Time Frame: Within 1 year after the study's Primary Completion Date (Last Subject Last Visit).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study included patients hospitalized with serious illness with laboratory-confirmed influenza A infection. Total 75 subjects were screened with 10 screen failures. Out of 65 randomized subjects, 60 received study treatment and 53 completed the study.
Groups:
- FLU-IGIV High Dose (450 mL): Participants received a single infusion of high dose of FLU-IGIV, administered over approximately 3 hours on Day 1. Administered intravenously at a dose of 450 mL of 65 g/mL FLU-IGIV diluted to 500 mL with normal saline. Participants also received standard of care (SOC) antiviral treatment for flu.
  FLU-IGIV: Single dose, sterile liquid formulation for IV administration.
- FLU-IGIV Low Dose (225 mL): Participants received a single infusion of low dose of FLU-IGIV, administered over approximately 3 hours on Day 1. Administered intravenously at a dose of 225 mL of 65 g/mL FLU-IGIV diluted to 500 mL with normal saline. Participants also received standard of care (SOC) antiviral treatment for flu.
  FLU-IGIV: Single dose, sterile liquid formulation for IV administration.
- Placebo (500 mL Normal Saline): Participants received a single infusion of placebo for FLU-IGIV, administered over approximately 3 hours on Day 1. Administered IV as 500 mL of normal saline. Participants also received SOC antiviral treatment for flu.
  Placebo for FLU-IGIV: Single dose, normal saline solution for IV administration.
Period: Overall Study
Arm/Group | FLU-IGIV High Dose (450 mL) | FLU-IGIV Low Dose (225 mL) | Placebo (500 mL Normal Saline)
Started | 21 | 20 | 24
Dosed (Safety Population) | 19 | 19 | 22
Completed | 18 | 16 | 19
Not Completed | 3 | 4 | 5

BASELINE CHARACTERISTICS:
Population: The ITT population includes all randomized subjects regardless of study medication (FLU-IGIV or placebo) dosing, influenza type or Protocol Deviations. Subjects are analyzed according to the treatment to which they were randomized. The ITT population is the primary analysis population for clinical benefit endpoints. Not all subjects had Day 8 data.
Groups:
- Total: Total of all reporting groups
Arm/Group | FLU-IGIV High Dose (450 mL) | FLU-IGIV Low Dose (225 mL) | Placebo (500 mL Normal Saline) | Total
Number analyzed (Participants) | 21 | 20 | 24 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (16.2) | 49.1 (14.2) | 59.5 (14.1) | 52.7 (15.5)
Age, Customized [Count of Participants; unit: Participants]
  18-54 | 13 | 11 | 8 | 32
  55 and over | 8 | 9 | 16 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 12 | 34
  Male | 9 | 10 | 12 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 3 | 10
  Not Hispanic or Latino | 18 | 16 | 21 | 55
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 9 | 14 | 32
  White | 12 | 11 | 10 | 33
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  North America | 20 | 20 | 22 | 62
  Spain | 1 | 0 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Frequency Counts and Percentage of Subjects With Adverse Events
Description: Frequency counts and percentage of subjects with Adverse Events by severity
Time Frame: Measured through Day 60
Population: The safety population includes all subjects who receive any amount of study medication (FLU-IGIV or placebo). In the case of incorrect treatment administration, subjects are analyzed according to the treatment received. The safety population is the primary analysis population for all safety data.
Measure: Count of Participants; unit: Participants
Arm/Group | FLU-IGIV High Dose (450 mL) | FLU-IGIV Low Dose (225 mL) | Placebo (500 mL Normal Saline)
Number analyzed (Participants) | 19 | 19 | 22
Participants
  Mild | 6 | 6 | 1
  Moderate | 3 | 5 | 6
  Severe | 1 | 1 | 4

2. Primary Outcome: Area Under the Plasma Concentration Curve [AUC] From Time 0 to 48 Hours Post-dose by Hemagglutinin Inhibition Assay
Description: Levels of anti-influenza A antibodies circulating in blood over time. We initially intended to look at this variable through Day 8, however, potential native antibody level changes and sparse sampling confounded results from 0 to 48 hours post-dose from PK samples collected from Baseline Day 1 pre-dose (time 0), Day 1 post-dose, Day 2 and Day 3 (if continued hospitalization), and Day 8. For AUC from time 0 to 48 hours, subjects who did not have a sample collected within +/-10% of 48 hours post-dose had this parameter set to missing, which is why the number of subjects who contributed data for this outcome measure is lower than the overall number of subjects analyzed.
Time Frame: Measured through 48 Hours post-dose
Population: The PK population includes all safety subjects who have adequate PK data for analysis that includes Day 1 baseline (pre-infusion) and at least one post-infusion time point. Subjects are analyzed according to the treatment received. See outcome measure description for subject exclusion details.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: titer*hours/mL
Arm/Group | FLU-IGIV High Dose (450 mL) | FLU-IGIV Low Dose (225 mL) | Placebo (500 mL Normal Saline)
Number analyzed (Participants) | 7 | 10 | 13
titer*hours/mL
  H1N1 California | 8589.9 (65.2) | 4955.4 (87.8) | 1973.1 (85.0)
  H1N1 Michigan | 5266.3 (67.6) | 3446.3 (123.2) | 1630.2 (106.4)
  H3N2 Hong Kong: number analyzed (Participants) | 7 | 10 | 11
  H3N2 Hong Kong | 11729.3 (47.4) | 7054.8 (39.1) | 3682.5 (126.7)
  H3N2 Singapore: number analyzed (Participants) | 7 | 10 | 11
  H3N2 Singapore | 6754.0 (34.2) | 4431.6 (45.3) | 2511.3 (219.6)

3. Primary Outcome: Maximum Plasma Concentration [Cmax] Reported as a Titer for Hemagglutinin Inhibition Assay
Description: Maximum observed concentration (reported as a titer) of anti-influenza A antibodies measured from Day 1 pre-dose (time 0) through Day 8 post-dose from PK samples collected from Baseline Day 1 pre-dose (time 0), Day 1 post-dose, Day 2 and Day 3 (if continued hospitalization), and Day 8.
Time Frame: Measured through Day 8 post-dose
Population: The PK population includes all safety subjects who have adequate PK data for analysis that includes Day 1 baseline (pre-infusion) and at least one post-infusion time point. Subjects are analyzed according to the treatment received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: titer
Arm/Group | FLU-IGIV High Dose (450 mL) | FLU-IGIV Low Dose (225 mL) | Placebo (500 mL Normal Saline)
Number analyzed (Participants) | 19 | 19 | 21
titer
  H1N1 California: number analyzed (Participants) | 19 | 19 | 20
  H1N1 California | 408.3 (99.8) | 152.5 (81.6) | 54.7 (135.9)
  H1N1 Michigan: number analyzed (Participants) | 19 | 19 | 18
  H1N1 Michigan | 371.6 (138.2) | 121.7 (114.6) | 54.7 (155.8)
  H3N2 Hong Kong: number analyzed (Participants) | 19 | 19 | 18
  H3N2 Hong Kong | 309.6 (38.4) | 239.8 (97.2) | 117.7 (317.2)
  H3N2 Singapore | 206.7 (35.1) | 192.7 (95.2) | 86.7 (297.0)

4. Primary Outcome: Time Cmax is Observed [Tmax] by Hemagglutinin Inhibition Assay
Description: Time that anti-influenza A antibodies are at maximum concentration from Day 1 pre-dose (time 0) through Day 8 post-dose from PK samples collected from Baseline Day 1 pre-dose (time 0), Day 1 post-dose, Day 2 and Day 3 (if continued hospitalization), and Day 8.
  The rate of study drug elimination and dependent parameters were not accurately estimable due to rising or sustained levels of anti-influenza A antibodies, this includes First Order Terminal Elimination Rate Constant [Kel], Plasma Clearance [Cl] and Total Volume of Distribution [Vz].
Time Frame: Measured through Day 8 post-dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | FLU-IGIV High Dose (450 mL) | FLU-IGIV Low Dose (225 mL) | Placebo (500 mL Normal Saline)
Number analyzed (Participants) | 19 | 19 | 21
hours
  H1N1 California: number analyzed (Participants) | 19 | 19 | 20
  H1N1 California | 24.4 (660.7) | 17.4 (358.8) | 108.7 (64.3)
  H1N1 Michigan: number analyzed (Participants) | 19 | 19 | 20
  H1N1 Michigan | 40.3 (522.5) | 13.9 (423.6) | 120.3 (58.4)
  H3N2 Hong Kong: number analyzed (Participants) | 19 | 19 | 18
  H3N2 Hong Kong | 4.8 (127.1) | 14.6 (298.4) | 76.8 (119.9)
  H3N2 Singapore: number analyzed (Participants) | 19 | 19 | 18
  H3N2 Singapore | 6.0 (146.0) | 23.0 (328.2) | 64.8 (171.4)

5. Secondary Outcome: Ordinal Scale Subject Distribution Reflecting Clinical Status
Description: Score (physician-assessed): 1=death; 2=hospitalization in the intensive care unit (ICU); 3=non-ICU hospitalization requiring supplemental oxygen; 4=non-ICU hospitalization not requiring supplemental oxygen; 5=no longer hospitalized but unable to resume normal activities; 6=no longer hospitalized with full resumption of normal activities. A higher score reflects improved clinical status. Not all ITT subjects had ordinal scale data available at Day 8 post-dose which explains why the overall number of participants analyzed is not consistent with the overall number of subjects included at baseline. For subjects who were discharged with unknown ordinal score the more conservative of two relevant discharged categories was imputed.
Time Frame: At Day 8 post-dose
Population: Intent to Treat (ITT) Population: includes all randomized subjects regardless of study medication (FLU-IGIV or placebo) dosing, influenza type or Protocol Deviations. Not all subjects had ordinal scale data available at Day 8 which is why the overall number of subjects analyzed is not consistent with the overall number of baseline subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | FLU-IGIV High Dose (450 mL) | FLU-IGIV Low Dose (225 mL) | Placebo (500 mL Normal Saline)
Number analyzed (Participants) | 19 | 17 | 21
Participants
  1-Death | 0 | 0 | 0
  2-Hospitalization in the ICU | 1 | 0 | 0
  3-Non-ICU hospitalization, requiring supp O2 | 0 | 2 | 4
  4-Non-ICU hospitalization, not requiring supp O2 | 0 | 0 | 0
  5-No longer hospitalized, no normal activities | 7 | 7 | 9
  6-No longer hospitalized, normal activities | 11 | 8 | 8
Statistical Analysis 1: Comparison: FLU-IGIV High Dose (450 mL) vs Placebo (500 mL Normal Saline); Pairwise Wilcoxon rank-sum test for a location shift; Test type: Superiority — A median estimated value of 0.000 indicates no difference between groups; p = 0.174, Wilcoxon (Mann-Whitney) — No adjustment for multiple comparisons, two-sided significance level of 0.05; Exact test; Median Difference (Net) = 0.000, 95.0% CI 2-sided [0.000 to 1.000] — FLU-IGIV High Dose (450 mL) - Placebo
Statistical Analysis 2: Comparison: FLU-IGIV Low Dose (225 mL) vs Placebo (500 mL Normal Saline); Pairwise Wilcoxon rank-sum test for a location shift; Test type: Superiority — A median estimated value of 0.000 indicates no difference between groups; p = 0.572, Wilcoxon (Mann-Whitney) — No adjustment for multiple comparisons, two-sided significance level of 0.05; Exact test; Mean Difference (Net) = 0.000, 95.0% CI 2-sided [0.000 to 1.000]
Statistical Analysis 3: Comparison: FLU-IGIV High Dose (450 mL) vs FLU-IGIV Low Dose (225 mL); Pairwise Wilcoxon rank-sum test for a location shift; Test type: Superiority — A median estimated value of 0.000 indicates no difference between groups; p = 0.534, Wilcoxon (Mann-Whitney) — No adjustment for multiple comparisons. two-sided significance level of 0.05; Exact test; Median Difference (Net) = 0.000, 95.0% CI 2-sided [0.000 to 1.000]
Statistical Analysis 4: Comparison: FLU-IGIV High Dose (450 mL) vs FLU-IGIV Low Dose (225 mL) vs Placebo (500 mL Normal Saline); Pairwise Wilcoxon rank-sum test for a location shift where the two active dose groups were pooled and compared to placebo; Test type: Superiority — A median estimated value of 0.000 indicates no difference between groups; p = 0.534, Wilcoxon (Mann-Whitney) — No adjustment for multiple comparisons, two-sided significance level of 0.05; Exact test; Median Difference (Net) = 0.000, 95.0% CI 2-sided [0.000 to 1.000] — FLU-IGIV pooled (450 mL + 250 mL) - Placebo

ADVERSE EVENTS:
Time Frame: From start of infusion on Day 1 through Day 60 (2 months).
Groups:
- Placebo (Normal Saline): Participants received a single infusion of placebo for FLU-IGIV, administered over approximately 3 hours on Day 1. Administered IV as 500 mL of normal saline. Participants also received SOC antiviral treatment for flu.
  Placebo for FLU-IGIV: Single dose, normal saline solution for IV administration.
Arm/Group | FLU-IGIV High Dose (450 mL) | FLU-IGIV Low Dose (225 mL) | Placebo (Normal Saline)
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19 | 0/22
Serious Adverse Events (participants affected / at risk) | 1/19 | 2/19 | 5/22
Other Adverse Events (participants affected / at risk) | 5/19 | 6/19 | 8/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FLU-IGIV High Dose (450 mL) (N=19) | FLU-IGIV Low Dose (225 mL) (N=19) | Placebo (Normal Saline) (N=22)
Cardiac Failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FLU-IGIV High Dose (450 mL) (N=19) | FLU-IGIV Low Dose (225 mL) (N=19) | Placebo (Normal Saline) (N=22)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Transaminases increased (Investigations) | 2 (2) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Physical deconditioning (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (3) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (2)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This phase 2 study was not powered to show efficacy. The target enrollment of 75 subjects randomized was not met (65 randomized and 60 dosed); the study was completed after the second northern hemisphere influenza season.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The result of the study may not be published until prior publication of the global results by the Sponsor, in the case of multi-center studies.

DOCUMENTS (2):
  • Study Protocol (2019-01-24): https://cdn.clinicaltrials.gov/large-docs/04/NCT03315104/Prot_001.pdf
  • Statistical Analysis Plan (2019-11-07): https://cdn.clinicaltrials.gov/large-docs/04/NCT03315104/SAP_000.pdf